CLINICAL TRIAL: NCT01157312
Title: Minimal Stimulation or Clomiphene Citrate as First Line Therapy in Women With Polycystic Ovary Syndrome
Brief Title: Minimal Stimulation or Clomiphene Citrate in Treatment of Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-290s; FMH-212-G
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; clomiphene citrate; minimal stimulation; infertility treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- minimal stimulation protocol (Experimental): 5 days of CC (100mg/day) from day 3 followed by 150 IU of highly purified uFSH on cycle day 9 for three treatment cycles
  Interventions: Drug: clomiphene citrate +highly purified uFSH
- clomiphene citrate(CC) (Active Comparator): 5 days of CC (100mg/day) from cycle day 3 for three treatment cycles.
  Interventions: Drug: clomiphene citrate

INTERVENTIONS:
Drug: clomiphene citrate +highly purified uFSH
  Arms: minimal stimulation protocol
Drug: clomiphene citrate
  Arms: clomiphene citrate(CC)

SUMMARY:
The purpose of this study is to compare and determine the the efficacy of minimal stimulation and clomiphene citrate(CC) as the first-line treatment in infertile women with Polycystic Ovary Syndrome(PCOS).

DETAILED DESCRIPTION:
All patients received 100 mg CC (Clomid®; Global Napi Pharmaceuticals, Cairo, Egypt) for 5 days starting from day 3 of spontaneous or induced menstruation. In group A (minimal stimulation), 2 vials of highly purified uFSH , 150 IU (Fostimon; IBSA, Lugano, Switzerland, 75 IU/vial) were given IM on cycle day 9. A total of 3 cycles was offered to each group.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* No other infertility factors
* No previous use of ovarian stimulation drugs

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing syndrome
* Androgen secreting tumors

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per cycle

SECONDARY OUTCOMES:
endometrial thickness at the time of hCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD MRCOG, Principal Investigator — Mansoura University Hospital; Mohamed F Bazeed, MD, Study Director — Mansoura University Hospital; Ibrahim Abd Elaal, MD, Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Lu PY, Chen AL, Atkinson EJ, Lee SH, Erickson LD, Ory SJ. Minimal stimulation achieves pregnancy rates comparable to human menopausal gonadotropins in the treatment of infertility. Fertil Steril. 1996 Mar;65(3):583-7. doi: 10.1016/s0015-0282(16)58158-8. PMID 8774291
- [Background] Houmard BS, Juang MP, Soules MR, Fujimoto VY. Factors influencing pregnancy rates with a combined clomiphene citrate/gonadotropin protocol for non-assisted reproductive technology fertility treatment. Fertil Steril. 2002 Feb;77(2):384-6. doi: 10.1016/s0015-0282(01)02990-9. PMID 11821101
- [Background] Dhaliwal LK, Sialy RK, Gopalan S, Majumdar S. Minimal stimulation protocol for use with intrauterine insemination in the treatment of infertility. J Obstet Gynaecol Res. 2002 Dec;28(6):295-9. doi: 10.1046/j.1341-8076.2002.00058.x. PMID 12512925
- [Derived] Abu Hashim H, Bazeed M, Abd Elaal I. Minimal stimulation or clomiphene citrate as first-line therapy in women with polycystic ovary syndrome: a randomized controlled trial. Gynecol Endocrinol. 2012 Feb;28(2):87-90. doi: 10.3109/09513590.2011.589924. Epub 2011 Jul 20. PMID 21770837